CLINICAL TRIAL: NCT05624515
Title: Efficacy of Dry Needling and Ischaemic Compression of the Scapula Angularis Muscle in Patients With Cervicalgia. Randomised Clinical Trial
Brief Title: Efficacy of Dry Needling in Cervical Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Principal Investigator, Universidad Católica de Ávila
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 14/11/2022
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Cervical Pain
Keywords: dry needling; physiotherapy techniques; cervical pain; pain
MeSH Terms: conditions — Neck Pain; Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dry needling group (Experimental): Subjects undergoing dry needling of the angularis scapulae muscle
  Interventions: Device: dry needling
- ischaemic compression group (Experimental): Subjects undergoing ischaemic compression of the angularis scapulae muscle
  Interventions: Other: Ischaemic compression

INTERVENTIONS:
Device: dry needling — Active trigger point puncture of the angularis scapulae muscle
  Arms: dry needling group
Other: Ischaemic compression — Ischaemic compression at the active trigger point of the angularis scapulae muscle
  Arms: ischaemic compression group

SUMMARY:
The presence of latent myofascial trigger points (MTrPs) in the angular muscle of the scapula is one of the possible causes of non-specific neck pain. Dry needling (DN) and ischaemic compression (IC) techniques may be useful for the treatment of these MTrPs. Methods: 80 participants were divided into two groups: the dry needling group, which received a single session of DN on the angular muscle plus hyperalgesia (n=40), and the IC group, which received a single session of IC on the angular muscle plus hyperalgesia (n=40). Pain intensity, pain pressure threshold (PPT), range of motion (ROM) and quality of life were assessed at baseline, immediately after, 48 hours and one week after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with neck pain
* Patients presenting with trigger point activation of the angularis scapulae muscle

Exclusion Criteria:

* Patients who have an absolute fear of needles (belonephobia).
* Patients presenting with cervical pain with radiculopathy or irradiation of pain to the upper limb.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 3 months
  Pain intensity measured on the VAS scale with a minimum score of 0 (no pain) and a maximum score of 10 (highest possible pain endured).

SECONDARY OUTCOMES:
pressure pain threshold | 3 months
  pressure on the sore spot measured by algometer and the unit is Newtons.
range of motion | 3 months
  Joint movement in the cervical spine measured in degrees using a goniometer
quality life | 3 months
  Measured by physical activity questionnaire. Scoring is based on patients' responses. Minimum of 0, maximum of 100 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica de Ávila, Ávila, Completado, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Navarro-Santana MJ, Sanchez-Infante J, Fernandez-de-Las-Penas C, Cleland JA, Martin-Casas P, Plaza-Manzano G. Effectiveness of Dry Needling for Myofascial Trigger Points Associated with Neck Pain Symptoms: An Updated Systematic Review and Meta-Analysis. J Clin Med. 2020 Oct 14;9(10):3300. doi: 10.3390/jcm9103300. PMID 33066556
- [Result] Ballyns JJ, Shah JP, Hammond J, Gebreab T, Gerber LH, Sikdar S. Objective sonographic measures for characterizing myofascial trigger points associated with cervical pain. J Ultrasound Med. 2011 Oct;30(10):1331-40. doi: 10.7863/jum.2011.30.10.1331. PMID 21968483
- [Result] Lluch E, Arguisuelas MD, Coloma PS, Palma F, Rey A, Falla D. Effects of deep cervical flexor training on pressure pain thresholds over myofascial trigger points in patients with chronic neck pain. J Manipulative Physiol Ther. 2013 Nov-Dec;36(9):604-11. doi: 10.1016/j.jmpt.2013.08.004. Epub 2013 Oct 21. PMID 24152997
- [Result] Lew J, Kim J, Nair P. Comparison of dry needling and trigger point manual therapy in patients with neck and upper back myofascial pain syndrome: a systematic review and meta-analysis. J Man Manip Ther. 2021 Jun;29(3):136-146. doi: 10.1080/10669817.2020.1822618. Epub 2020 Sep 22. PMID 32962567
- [Result] Kietrys DM, Palombaro KM, Azzaretto E, Hubler R, Schaller B, Schlussel JM, Tucker M. Effectiveness of dry needling for upper-quarter myofascial pain: a systematic review and meta-analysis. J Orthop Sports Phys Ther. 2013 Sep;43(9):620-34. doi: 10.2519/jospt.2013.4668. PMID 23756457
- [Result] Stieven FF, Ferreira GE, de Araujo FX, Angellos RF, Silva MF, da Rosa LHT. Immediate Effects of Dry Needling and Myofascial Release on Local and Widespread Pressure Pain Threshold in Individuals With Active Upper Trapezius Trigger Points: A Randomized Clinical Trial. J Manipulative Physiol Ther. 2021 Feb;44(2):95-102. doi: 10.1016/j.jmpt.2020.07.003. Epub 2021 Jan 9. PMID 33431282